CLINICAL TRIAL: NCT04369287
Title: Prevalence, Correlation With Other Mutant Genes and Clinical Effect of IDH1/2 Mutations in Patients With Acute Myeloid Leukemia. The European IDH Research Alliance
Brief Title: Prevalence and Clinical Effect of IDH1/2 Mutations in Patients With Acute Myeloid Leukemia
Acronym: Euro_IDH_AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC/OSS-04/2016
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Acute Myeloid Leukemia; IDH1 Gene Mutation; IDH2 Gene Mutation
Keywords: AML, IDH1 gene, IDH2 gene, gene mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood (PB) and bone marrow (BM) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IDH1-mutated AML: Patients affected with AML and carryng IDH1 mutations
- IDH2-mutated AML: Patients affected with AML and carryng IDH2 mutations
- IDH1/2 unmutated AML: Patients affected with AML without IDH1/2 mutations

SUMMARY:
Among the most notable cancer genome-wide sequencing discoveries in recent years was the finding of mutation hot-spots in the isocitrate dehydrogenase (IDH) genes in grade II/III astrocytomas and oligodendrogliomas and in secondary glioblastomas. This was rapidly followed by identification of recurrent IDH1/2 mutations in myeloid neoplasms (MN), including acute myeloid leukemia (AML). Mutant IDH is now a therapeutic target of great interest in cancer research, especially in AML, given the limitations of current approved therapies and the encouraging early clinical data demonstrating proof of concept for investigational mutant IDH1/2 inhibitors.

The origin of mutations in AML was explored by investigating the clonal evolution of genomes sequenced from patients with M1- or M3-AML and comparing them with hematopoietic stem/progenitor cells (HSPCs) from healthy volunteers. Six genes were found to have statistically higher mutation frequencies in M1 versus M3 genomes (NPM1, DNMT3A, IDH1, IDH2, TET2 and ASXL1), suggesting they are initiating rather than cooperating events. Prospective evaluation of serial 2- HG levels during treatment of newly diagnosed AML treated with standard chemotherapy revealed that both 2-HG level and mutated IDH allele burden decreased with response to treatment but began to rise again as therapy failed.

The prognostic impact of IDH mutations in AML is under continued investigation and varies across studies. In this research project authors aim a) to define the prevalence and type of IDH1/2 mutations in AML patients; b) to define relationships between IDH1/2 mutations and other oncogenic mutations in AML, as well as to describe clonal evolution of the disease and c) to describe the clinical outcome of IDH1/2 mutated patients with AML treated with currently available treatments.

DETAILED DESCRIPTION:
Among the most notable cancer genome-wide sequencing discoveries in recent years was the finding of mutation hot-spots in the isocitrate dehydrogenase (IDH) genes in grade II/III astrocytomas and oligodendrogliomas and in secondary glioblastomas. This was rapidly followed by identification of recurrent IDH1/2 mutations in myeloid neoplasms (MN), including acute myeloid leukemia (AML), myelodysplastic syndromes (MDS) and myeloproliferative neoplasms (MPN).

Mutant IDH is now a therapeutic target of great interest in cancer research, especially in AML, given the limitations of current approved therapies and the encouraging early clinical data demonstrating proof of concept for investigational mutant IDH1/2 inhibitors.

There is evidence to suggest that IDH mutations may cooperate with other mutations to initiate and drive oncogenesis in myeloid malignancies. High levels of 2-hydroxyglutarate (2-HG, as a result of gene mutation) have been shown to inhibit αKG-dependent dioxygenases including histone and DNA demethylases, proteins that regulate cellular epigenetic status. Consistent with 2-HG promoting cancer via an effect on chromatin structure, tumors harboring IDH mutations display a CpG island methylator phenotype. More recent studies have shown that overexpression of mutant IDH enzymes can induce histone and DNA hypermethylation, as well as block cellular differentiation. Together, these data suggest that cancer-associated IDH mutations can induce a block in cellular differentiation through epigenetic modifications, which contributes to tumor initiation and progression, and thus support the clinical evaluation of agents targeted to mutant IDH

The origin of mutations in AML was explored by investigating the clonal evolution of genomes sequenced from patients with M1- or M3-AML and comparing them with hematopoietic stem/progenitor cells (HSPCs) from healthy volunteers. Six genes were found to have statistically higher mutation frequencies in M1 versus M3 genomes (NPM1, DNMT3A, IDH1, IDH2, TET2 and ASXL1), suggesting they are initiating rather than cooperating events. Furthermore, all of these genes have been shown to play a role in chromatin modification, suggesting that epigenetic alterations may function to initiate tumorigenesis.

Prospective evaluation of serial 2-HG levels during treatment of newly diagnosed AML treated with standard chemotherapy revealed that both 2-HG level and mutated IDH allele burden decreased with response to treatment but began to rise again as therapy failed.

The prognostic impact of IDH mutations in AML is under continued investigation and varies across studies

In this research project, the authors aim:

1. To define the prevalence and type of IDH1/2 mutations in acute myeloid leukemias.
2. To define genotype-phenotype relationship in IDH1/2 mutated patients.
3. To define relationships between IDH1/2 mutations and other oncogenic mutations in AML, as well as to describe clonal evolution of the disease (including the evaluation of genotype at disease relapse).
4. To describe the clinical outcome of IDH1/2 mutated patients with AML treated with currently available treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of AML According to 2016 WHO classification criteria
* Ability to give informed consent according to ICH/EU GCP, and national/local regulations.

Exclusion Criteria:

* Lack of written informed consent
* Lack of biological samples (blood, bone marrow aspirate)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IDH 1/2 mutated patients, IDH not mutaded patients
Sampling Method: Non-Probability Sample
Enrollment: 654 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of IDH1/2 mutations in patients with AML | 2016-2020
  IDH1/2 mutational status will be analyzed in all centers by NGS or sanger sequencing on samples obtained from patients affected with AML enrolled in the study with the aim to provide information on the prevalence and type of IDH1/2 mutations
genotype-phenotype correlations in AML patients carryng IDH1/2 mutations | 2016-2020
  Data obtained from targeted gene sequencing will be correlated with clinical and hematological variables of interest (i.e., demographic factors, WHO 2016 category, cytogenetics, presence of recurrent molecular abnormalities, response to treatment, overall survival, disease-free survival) to identify specific associations between genotype and disease phenotype)
Overall survival in patients with AML carryng IDH1/2 mutations | 2016-2020
  Specific analyses will be carried out to describe overall survival of AML with IDH1/2 mutations with currently available treatments. Moreover, A comparison between survival of IDH-mutated vs. IDH-unmutated patients will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Sole, MD, Principal Investigator — Josep Carreras Leukaemia Research Institute; Joana Desterro, Principal Investigator — Instituto Português de Oncologia de Lisboa; Klaus Metzeler, Principal Investigator — Laboratory for Leukemia Diagnostics. University of Munich; Pau Montesinos, Principal Investigator — Hematology Department. Hospital Universitari i Politècnic La Fe; Jorge Sierra, Principal Investigator — Hospital de la Santa Creu i Sant Pau Autonomous University of Barcelona, Spain; Matteo Della Porta, MD, Study Chair — Humanitas Research Hospital IRCCS, Rozzano-Milan; Maria Teresa Voso, Principal Investigator — Fondazione GIMEMA; Christoph Roellig, Principal Investigator — Technische Universität Dresden | TUD · Medical Clinic; Lisa Pleyer, Principal Investigator — Salzburg Cancer Reasearch Institute (SCRI), Cancer Cluster Salzburg (CCS); Moritz Middeke, Principal Investigator — Technische Universität Dresden | TUD · Medical Clinic
Locations (1):
- Istituto Clinico Humanitas, Milan, Italy

REFERENCES:
- [Result] Larsson CA, Cote G, Quintas-Cardama A. The changing mutational landscape of acute myeloid leukemia and myelodysplastic syndrome. Mol Cancer Res. 2013 Aug;11(8):815-27. doi: 10.1158/1541-7786.MCR-12-0695. Epub 2013 May 3. PMID 23645565
- [Result] Chou WC, Lei WC, Ko BS, Hou HA, Chen CY, Tang JL, Yao M, Tsay W, Wu SJ, Huang SY, Hsu SC, Chen YC, Chang YC, Kuo KT, Lee FY, Liu MC, Liu CW, Tseng MH, Huang CF, Tien HF. The prognostic impact and stability of Isocitrate dehydrogenase 2 mutation in adult patients with acute myeloid leukemia. Leukemia. 2011 Feb;25(2):246-53. doi: 10.1038/leu.2010.267. Epub 2010 Nov 16. PMID 21079611
- [Result] DiNardo CD, Ravandi F, Agresta S, Konopleva M, Takahashi K, Kadia T, Routbort M, Patel KP, Mark Brandt, Pierce S, Garcia-Manero G, Cortes J, Kantarjian H. Characteristics, clinical outcome, and prognostic significance of IDH mutations in AML. Am J Hematol. 2015 Aug;90(8):732-6. doi: 10.1002/ajh.24072. PMID 26016821
- [Result] Thol F, Damm F, Wagner K, Gohring G, Schlegelberger B, Hoelzer D, Lubbert M, Heit W, Kanz L, Schlimok G, Raghavachar A, Fiedler W, Kirchner H, Heil G, Heuser M, Krauter J, Ganser A. Prognostic impact of IDH2 mutations in cytogenetically normal acute myeloid leukemia. Blood. 2010 Jul 29;116(4):614-6. doi: 10.1182/blood-2010-03-272146. Epub 2010 Apr 26. PMID 20421455
- [Result] Cancer Genome Atlas Research Network; Ley TJ, Miller C, Ding L, Raphael BJ, Mungall AJ, Robertson A, Hoadley K, Triche TJ Jr, Laird PW, Baty JD, Fulton LL, Fulton R, Heath SE, Kalicki-Veizer J, Kandoth C, Klco JM, Koboldt DC, Kanchi KL, Kulkarni S, Lamprecht TL, Larson DE, Lin L, Lu C, McLellan MD, McMichael JF, Payton J, Schmidt H, Spencer DH, Tomasson MH, Wallis JW, Wartman LD, Watson MA, Welch J, Wendl MC, Ally A, Balasundaram M, Birol I, Butterfield Y, Chiu R, Chu A, Chuah E, Chun HJ, Corbett R, Dhalla N, Guin R, He A, Hirst C, Hirst M, Holt RA, Jones S, Karsan A, Lee D, Li HI, Marra MA, Mayo M, Moore RA, Mungall K, Parker J, Pleasance E, Plettner P, Schein J, Stoll D, Swanson L, Tam A, Thiessen N, Varhol R, Wye N, Zhao Y, Gabriel S, Getz G, Sougnez C, Zou L, Leiserson MD, Vandin F, Wu HT, Applebaum F, Baylin SB, Akbani R, Broom BM, Chen K, Motter TC, Nguyen K, Weinstein JN, Zhang N, Ferguson ML, Adams C, Black A, Bowen J, Gastier-Foster J, Grossman T, Lichtenberg T, Wise L, Davidsen T, Demchok JA, Shaw KR, Sheth M, Sofia HJ, Yang L, Downing JR, Eley G. Genomic and epigenomic landscapes of adult de novo acute myeloid leukemia. N Engl J Med. 2013 May 30;368(22):2059-74. doi: 10.1056/NEJMoa1301689. Epub 2013 May 1. PMID 23634996
- [Result] Papaemmanuil E, Gerstung M, Malcovati L, Tauro S, Gundem G, Van Loo P, Yoon CJ, Ellis P, Wedge DC, Pellagatti A, Shlien A, Groves MJ, Forbes SA, Raine K, Hinton J, Mudie LJ, McLaren S, Hardy C, Latimer C, Della Porta MG, O'Meara S, Ambaglio I, Galli A, Butler AP, Walldin G, Teague JW, Quek L, Sternberg A, Gambacorti-Passerini C, Cross NC, Green AR, Boultwood J, Vyas P, Hellstrom-Lindberg E, Bowen D, Cazzola M, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Clinical and biological implications of driver mutations in myelodysplastic syndromes. Blood. 2013 Nov 21;122(22):3616-27; quiz 3699. doi: 10.1182/blood-2013-08-518886. Epub 2013 Sep 12. PMID 24030381
- [Result] Ward PS, Patel J, Wise DR, Abdel-Wahab O, Bennett BD, Coller HA, Cross JR, Fantin VR, Hedvat CV, Perl AE, Rabinowitz JD, Carroll M, Su SM, Sharp KA, Levine RL, Thompson CB. The common feature of leukemia-associated IDH1 and IDH2 mutations is a neomorphic enzyme activity converting alpha-ketoglutarate to 2-hydroxyglutarate. Cancer Cell. 2010 Mar 16;17(3):225-34. doi: 10.1016/j.ccr.2010.01.020. Epub 2010 Feb 18. PMID 20171147
- [Result] Gross S, Cairns RA, Minden MD, Driggers EM, Bittinger MA, Jang HG, Sasaki M, Jin S, Schenkein DP, Su SM, Dang L, Fantin VR, Mak TW. Cancer-associated metabolite 2-hydroxyglutarate accumulates in acute myelogenous leukemia with isocitrate dehydrogenase 1 and 2 mutations. J Exp Med. 2010 Feb 15;207(2):339-44. doi: 10.1084/jem.20092506. Epub 2010 Feb 8. PMID 20142433
- [Result] DiNardo CD, Propert KJ, Loren AW, Paietta E, Sun Z, Levine RL, Straley KS, Yen K, Patel JP, Agresta S, Abdel-Wahab O, Perl AE, Litzow MR, Rowe JM, Lazarus HM, Fernandez HF, Margolis DJ, Tallman MS, Luger SM, Carroll M. Serum 2-hydroxyglutarate levels predict isocitrate dehydrogenase mutations and clinical outcome in acute myeloid leukemia. Blood. 2013 Jun 13;121(24):4917-24. doi: 10.1182/blood-2013-03-493197. Epub 2013 May 2. PMID 23641016
- [Result] Figueroa ME, Abdel-Wahab O, Lu C, Ward PS, Patel J, Shih A, Li Y, Bhagwat N, Vasanthakumar A, Fernandez HF, Tallman MS, Sun Z, Wolniak K, Peeters JK, Liu W, Choe SE, Fantin VR, Paietta E, Lowenberg B, Licht JD, Godley LA, Delwel R, Valk PJ, Thompson CB, Levine RL, Melnick A. Leukemic IDH1 and IDH2 mutations result in a hypermethylation phenotype, disrupt TET2 function, and impair hematopoietic differentiation. Cancer Cell. 2010 Dec 14;18(6):553-67. doi: 10.1016/j.ccr.2010.11.015. Epub 2010 Dec 9. PMID 21130701
- [Result] Ye D, Xiong Y, Guan KL. The mechanisms of IDH mutations in tumorigenesis. Cell Res. 2012 Jul;22(7):1102-4. doi: 10.1038/cr.2012.51. Epub 2012 Mar 27. PMID 22453240
- [Result] Wang F, Travins J, DeLaBarre B, Penard-Lacronique V, Schalm S, Hansen E, Straley K, Kernytsky A, Liu W, Gliser C, Yang H, Gross S, Artin E, Saada V, Mylonas E, Quivoron C, Popovici-Muller J, Saunders JO, Salituro FG, Yan S, Murray S, Wei W, Gao Y, Dang L, Dorsch M, Agresta S, Schenkein DP, Biller SA, Su SM, de Botton S, Yen KE. Targeted inhibition of mutant IDH2 in leukemia cells induces cellular differentiation. Science. 2013 May 3;340(6132):622-6. doi: 10.1126/science.1234769. Epub 2013 Apr 4. PMID 23558173
- [Result] Losman JA, Looper RE, Koivunen P, Lee S, Schneider RK, McMahon C, Cowley GS, Root DE, Ebert BL, Kaelin WG Jr. (R)-2-hydroxyglutarate is sufficient to promote leukemogenesis and its effects are reversible. Science. 2013 Mar 29;339(6127):1621-5. doi: 10.1126/science.1231677. Epub 2013 Feb 7. PMID 23393090
- [Result] Della Porta MG, Travaglino E, Boveri E, Ponzoni M, Malcovati L, Papaemmanuil E, Rigolin GM, Pascutto C, Croci G, Gianelli U, Milani R, Ambaglio I, Elena C, Ubezio M, Da Via' MC, Bono E, Pietra D, Quaglia F, Bastia R, Ferretti V, Cuneo A, Morra E, Campbell PJ, Orazi A, Invernizzi R, Cazzola M; Rete Ematologica Lombarda (REL) Clinical Network. Minimal morphological criteria for defining bone marrow dysplasia: a basis for clinical implementation of WHO classification of myelodysplastic syndromes. Leukemia. 2015 Jan;29(1):66-75. doi: 10.1038/leu.2014.161. Epub 2014 May 20. PMID 24935723